CLINICAL TRIAL: NCT04441736
Title: Different Oxygenation Modalities for Early Post Extubation Failure
Brief Title: Post -Extubation Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Farouk, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MS-313-2019
Record Dates: First submitted 2020-06-10; First posted 2020-06-22 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High flow nasal cannula (Active Comparator): A device of high flow nasal cannula giving 60 litres / min flow
  Interventions: Device: High flow nasal cannula
- Conventional oxygen (Placebo Comparator): Nasal cannula giving oxygen up to 10 litres / minute
  Interventions: Device: High flow nasal cannula
- Non invasive ventilation (Active Comparator): non invasive ventilation with IPAP and EPAP
  Interventions: Device: High flow nasal cannula

INTERVENTIONS:
Device: High flow nasal cannula — Device gives high flow oxygen comparable to non invasive ventilation and conventional oxygen therapy
  Other Names: Non invasive ventilation

SUMMARY:
comparing high flow nasal cannula , conventional oxygen tharapy and non invasive ventilation post-extubation period for patients mechanically ventilated due to respiratory failure regarding re-intubation rate, ICU outcome & 28 days mortality

DETAILED DESCRIPTION:
patients with respiratory failure either type I or type II planned for extubation will be divided into 3 groups post extubation :

Group I: will receive high flow nasal cannula giving oxygen 60 litres / minute flow group II: will receive nasal cannula up to 10 litres / minute group III: will receive non invasive ventilation

Data of the patients will be collected for 28 days post-extubation and analysed

ELIGIBILITY:
Inclusion Criteria:

* respiratory failure type I and Type II

Exclusion Criteria:

* Mechanical ventilation due to other cause such as disturbed conscious level or respiratory muscle weakness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with post extubation respiratory failure | 7 days
  Number of participants with post extubation hypoxemia with or without hypercapnea

SECONDARY OUTCOMES:
Rate of ICU stay and mortality | 28 days
  Duration of ICU stay and incidence of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Nassar, MD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No